CLINICAL TRIAL: NCT05708157
Title: Therapeutic Role of Concomitant Intranasal Antihistamine and Corticosteroid in Patient With Perennial Allergic Rhinitis Whose Symptoms Are Not Controlled With Intranasal Corticosteroid
Brief Title: Concomitant Intranasal Antihistamine and Corticosteroid in Stepwise Treatment Strategy for Allergic Rhinitis
Acronym: INCS/INAH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Hallym University Kangnam Sacred Heart Hospital (Other); Gangneung Asan Hospital (Other); Bundang Jesaeng Hospital (Unknown); Chung-Ang University Gwangmyeong Hospital (Other); Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Sangmin Lee, MD, Professor, Gachon University Gil Medical Center
Other Study IDs: GCIRB2022-327
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active group: Patients with perennial allergic rhinitis who receive concomitant intranasal antihistamine and corticosteroid.
  Interventions: Drug: concomitant intranasal antihistamine and corticosteroid

INTERVENTIONS:
Drug: concomitant intranasal antihistamine and corticosteroid — concomitant intranasal administration with antihistamine and corticosteroid

SUMMARY:
Patients with perennial allergic rhinitis whose symptoms are not controlled (visual analogue scale [VAS] ≥5) by 2-week treatment with intranasal corticosteroid will receive concomitant intranasal antihistamine and corticosteroid for 2 weeks. After 2-week treatment, changes in clinical parameters including VAS, total nasal symptom score (TNSS), total ocular symptom score (TOSS), rhinoconjunctivitis quality-of-life questionnaires (RQLQ) will be evaluated.

DETAILED DESCRIPTION:
Patients with perennial allergic rhinitis whose symptoms are not controlled (visual analogue scale [VAS] ≥5) by 2-week treatment with intranasal corticosteroid will receive concomitant intranasal antihistamine and corticosteroid. In addition to VAS, total nasal symptom score (TNSS), total ocular symptom score (TOSS), rhinoconjunctivitis quality-of-life questionnaires (RQLQ) will be measured before treatment (baseline) and 2 week after treatment. The differences between parameters before treatment and those after 2-week treatment will be statistically analyzed using paired student t test, and p<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Perinnial allergic rhinitis diagnosed by a doctor
* Positive for one or more of inhalant perinneal allergen in skin prick test or serum specific IgE measurement
* Age: 19 years or older
* Allergic rhinitis symptoms not controlled (VAS ≥5) by 2-week treatment with intranasal corticosteroid

Exclusion Criteria:

* Compliance for one or more drugs in last 2 weeks: <80%
* Use of oral corticosteroid, oral or intranasal decongestant in last 2 weeks
* Initiation of allergen-specific immunotherapy in last 12 months
* Seasonal allergic rhinitis
* Chronic rhinosinusitis other than allergic rhinitis
* Nasal polyposis
* Comorbid diseases including infectious, respiratory, cardiologic, renal, gastrointestinal, endocrinologic, oncologic, hemotologic and immunologic disorders which investigators judge to affect on the study significantly.
* Patients' rejection
* Pregenancy or lactation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with perennial allergic rhinitis whose symptoms are not controlled by 2-week treatement with intranasal corticosteroid.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
TNSS | 2 week
  total nasal symptom score

SECONDARY OUTCOMES:
TOSS | 2 week
  total nasal symptom score
RQLQ | 2 week
  rhinoconjunctivitis quality-of-life questionnares
VAS | 2 week
  visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Sang Min Lee, MD, PhD, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim M, Ryu G, Kang SY, Kim MA, Yang SI, Lee IH, Choi GS, Kim HJ, Lee SM, Kim DK, Choi JH, Yang HJ, Kim SW; Work Group for Rhinitis, the Korean Academy of Asthma, Allergy and Clinical Immunology. Intranasal antihistamine and corticosteroid to treat allergic rhinitis: A systematic review and meta-analysis. Allergy. 2022 Nov;77(11):3436-3440. doi: 10.1111/all.15415. Epub 2022 Jul 8. No abstract available. PMID 35716356